CLINICAL TRIAL: NCT00005330
Title: Framingham Children's Study - Food and Exercise Habits in Framingham Study Descendents
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4148; R01HL035653 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To identify early childhood determinants of eating and exercise behaviors that relate to cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

While dietary and physical activity habits are known to relate to cardiovascular risk, in 1985 little data were available on factors that influence the development of such behaviors early in life. In 1987, 106 families with 3 to 5 year old children were recruited to take part in the Framingham Children's Study. The children and their parents are direct descendents (4th and 3rd generation, respectively) of participants in the Framingham Heart Study. During the initial grant period, the feasibility of collecting relevant data has been demonstrated. Maintenance of the cohort and acceptance of the monitoring procedures have been excellent, due partly to the fact that the families consider themselves a part of the Framingham Heart Study and take pride in long-term compliance with study procedures.

DESIGN NARRATIVE:

The investigators have been following 100 families who are 3rd and 4th generation descendants of the original Framingham Heart Study cohort. The subjects were age 3-5 years at the onset of the study and were ages 11-14 years in 1996. There has been excellent cohort maintenance with over 90 percent of the original families continuing to participate. The study was renewed in FY 1996 to extend the Framingham Children's Study (FCS) to permit the evaluation of the determinants of change in the child's risk behaviors and other risk factors from early childhood through puberty to mid to late teens, a time when the individual's risk profile should better reflect his/her cardiovascular risk status as an adult.

The FCS is a longitudinal source of data on diet, activity and family and environmental factors in children. By 1996, the investigators had collected extensive dietary data with an average of 32 days of diet records and almost 50 days of electronically monitored physical activity data for each subject. Additional data included psychosocial and anthropometric data on children and their parents. The extension of the FCS allows continued monitoring of eating behaviors and physical activity habits of the children and their parents, as well as the personal environmental and behavioral factors influencing changes in the child's physical activity, diet, blood pressure, lipids and obesity from pre-school into the late teen years.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-09; Study Completion 2001-04 (Actual)

REFERENCES:
- [Background] Oliveria SA, Ellison RC, Moore LL, Gillman MW, Garrahie EJ, Singer MR. Parent-child relationships in nutrient intake: the Framingham Children's Study. Am J Clin Nutr. 1992 Sep;56(3):593-8. doi: 10.1093/ajcn/56.3.593. PMID 1503074
- [Background] Gillman MW, Cupples LA, Moore LL, Ellison RC. Impact of within-person variability on identifying children with hypercholesterolemia: Framingham Children's Study. J Pediatr. 1992 Sep;121(3):342-7. doi: 10.1016/s0022-3476(05)81785-8. PMID 1517906
- [Background] Gillman MW, Oliveria SA, Moore LL, Ellison RC. Inverse association of dietary calcium with systolic blood pressure in young children. JAMA. 1992 May 6;267(17):2340-3. PMID 1564773
- [Background] Garrahie EJ, Humphrey KF, Witschi JC, Stephenson WP, Ellison RC. The value of debriefing mothers of 3- to 7-year-old children when analyzing children's food diaries. J Am Diet Assoc. 1991 Jun;91(6):710-1. No abstract available. PMID 2040786
- [Background] Marmor JK, Oliveria SA, Donahue RP, Garrahie EJ, White MJ, Moore LL, Ellison RC. Factors encouraging cohort maintenance in a longitudinal study. J Clin Epidemiol. 1991;44(6):531-5. doi: 10.1016/0895-4356(91)90216-v. PMID 2037857
- [Background] Moore LL, Lombardi DA, White MJ, Campbell JL, Oliveria SA, Ellison RC. Influence of parents' physical activity levels on activity levels of young children. J Pediatr. 1991 Feb;118(2):215-9. doi: 10.1016/s0022-3476(05)80485-8. PMID 1993947
- [Background] Ellison RC, Singer MR, Moore LL, Nguyen US, Garrahie EJ, Marmor JK. Current caffeine intake of young children: amount and sources. J Am Diet Assoc. 1995 Jul;95(7):802-4. doi: 10.1016/S0002-8223(95)00222-7. No abstract available. PMID 7797813
- [Background] Singer MR, Moore LL, Garrahie EJ, Ellison RC. The tracking of nutrient intake in young children: the Framingham Children's Study. Am J Public Health. 1995 Dec;85(12):1673-7. doi: 10.2105/ajph.85.12.1673. PMID 7503343
- [Background] Moore LL, Nguyen US, Rothman KJ, Cupples LA, Ellison RC. Preschool physical activity level and change in body fatness in young children. The Framingham Children's Study. Am J Epidemiol. 1995 Nov 1;142(9):982-8. doi: 10.1093/oxfordjournals.aje.a117747. PMID 7572980
- [Background] Hood MY, Moore LL, Sundarajan-Ramamurti A, Singer M, Cupples LA, Ellison RC. Parental eating attitudes and the development of obesity in children. The Framingham Children's Study. Int J Obes Relat Metab Disord. 2000 Oct;24(10):1319-25. doi: 10.1038/sj.ijo.0801396. PMID 11093294